CLINICAL TRIAL: NCT02768441
Title: Pharmacokinetics of New Dexamphetamine Sustained Release Tablets and the Clinical Validation of Measuring Dexamphetamine in Dried Blood Spots
Brief Title: Dexamphetamine Sustained Release Pharmacokinetics and Clinical Validation of Dried Blood Spots
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAM001DFM
Record Dates: First submitted 2016-04-26; First posted 2016-05-11 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Cocaine Addiction
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Dextroamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): Participants receiving Dexamphetamine 60 mg SR
  Interventions: Drug: Dexamphetamine

INTERVENTIONS:
Drug: Dexamphetamine — Participants will receive 60 mg Dexamphetamine SR daily for 5 consecutive days

SUMMARY:
The pharmacokinetics of 10 to 12 individuals receiving 60 mg of sustained release dexamphetamine will be studied. These individuals have received this medication before in a previous trial where the pharmacodynamics were investigated. This trial will last 5 consecutive days during which blood samples will be drawn for pharmacokinetics analyses. Dried blood spots will also be collected for the clinical validation of the bioanalytical method wherein these are used.

ELIGIBILITY:
Inclusion Criteria:

* Have completed at least 80% of the previous study (CATCH)
* Be able and willing to participate in the study and assessments
* Have provided written informed consent.

Exclusion Criteria:

* Any intake of dexamphetamine 7 days or less before the start of the proposed study;
* Contraindications for dexamphetamine
* (desired) pregnancy or continued lactation
* Insufficient command of the Dutch language
* Current participation in another trial

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (AUC) of dexamphetamine | Determined on the 5 day bloodsamples taken
Maximum plasma concentration (Cmax) of dexamphetamine | Determined on the 5 day bloodsamples taken
Half life (T 1/2) of dexamphetamine | Determined on the 5 day bloodsamples taken

CONTACTS AND LOCATIONS:
Overall Officials: Wim van den Brink, PhD, Principal Investigator — Academic Psychiatric Center AMC-UvA
Locations (1):
- AMC, Amsterdam, Netherlands